CLINICAL TRIAL: NCT03328559
Title: Kinetics of Circulating Tumoral Cells in Bronchial Primitive Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTC
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Bronchial Cancer
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early stage bronchial cancer (Other): Early stage which can benefit from a surgical resection. A taking will be made in preoperative then in every consultation of follow-up after the intervention
  Interventions: Diagnostic Test: ISET® - Isolation by Size of Tumor cells
- advanced stage bronchial cancer (Other): Patients locally moved forward or at a metastatic stage handled by chemotherapy
  Interventions: Diagnostic Test: ISET® - Isolation by Size of Tumor cells

INTERVENTIONS:
Diagnostic Test: ISET® - Isolation by Size of Tumor cells — early stage bronchial cancer patient will have a blood collection
  Arms: early stage bronchial cancer
Diagnostic Test: ISET® - Isolation by Size of Tumor cells — advanced stage bronchial cancer patient will have a blood collection
  Arms: advanced stage bronchial cancer

SUMMARY:
The pronostic value of Circulating Tumoral Cells(CTC) 's dosage by the method ISET® (tumoral cell isolation by size) in patients with bronchial cancer was previously demonstrated.

However, no kinetic study was ever realized to study the value of the CTC as predictive indicator of answer to the therapy. This project plans to study patients in an early stage and patients at advance stage locally moved forward or metastatic of the disease by evaluation of the presence and the number of CTC before every cure. This collaborative and original study should allow to refine the diagnoses of answer and to plan the possible relapses what would allow a premature institution of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-small cell lung cancer
* accepting participation

Exclusion Criteria:

* refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
numeration of CTC (circulant tumoral cell) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean P Tredaniel, Pr, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France